CLINICAL TRIAL: NCT05518838
Title: Expanded Access to OKN-007 for Patients With Diffuse Midline Glioma, H3 K27-altered
Status: No longer available | Type: Expanded Access
Sponsor: Oblato, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: OKN-007-EA-DMG
Record Dates: First submitted 2022-08-24; First posted 2022-08-29 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Diffuse Midline Glioma, H3 K27M-Mutant; Diffuse Intrinsic Pontine Glioma
MeSH Terms: conditions — Diffuse Intrinsic Pontine Glioma | interventions — OKN 007

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: OKN-007 — OKN-007 is an intravenously administrated drug being developed as a novel anti-cancer therapy against gliomas.

SUMMARY:
To provide OKN-007 for compassionate use in patients with diffuse midline glioma, H3 K27-altered (DMG), including diffuse intrinsic pontine glioma (DIPG), pediatric and young adult patients with high-grade diffuse midline glioma will be treated under this Intermediate-sized expanded access treatment protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Age from > 12 months to ≤ 18 years of age at the time of enrollment.
2. Diagnosis of diffuse midline glioma, H3 K27-altered according to the WHO 2021 Classification of Tumors of the Central Nervous System diagnostic criteria including diffuse intrinsic pontine glioma (DIPG). In the absence of a pathologically confirmed diagnosis, a grade IV glioma involving the thalamus, hypothalamus, brainstem, cerebellum, midbrain, or spinal cord, or with a pontine epicenter and diffuse involvement of the pons.
3. Patient has completed definitive radiation therapy as part of standard-of-care treatment or was unable to undergo radiation.
4. Karnofsky performance status ≥ 50 for patients ≥ 16 years of age and Lansky performance status ≥ 50 for patients < 16 years of age; patients who are unable to walk because of paralysis, but who are upright in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
5. Patients must have adequate bone marrow, liver, and renal function:
6. For females of childbearing potential, negative urinary or serum pregnancy test.
7. Patients must be willing to highly effective contraception for both male and female patients throughout the treatment and for at least 4 months after last treatment administration.
8. Toxicities related to any prior treatments are either stable, stable on supportive therapy, resolved, or in the opinion of the treating physician, clinically non-significant
9. Ability to understand a written informed consent document, and the willingness to sign it. Assent will be obtained when appropriate based on the patient's age.

Exclusion Criteria:

1. Patient is already participating in or qualifies for and is able to enroll in a clinical trial of OKN-007 and other ongoing clinical trials.
2. Patient has received systemic therapy with an investigational agent within 5 half-lives or 14 days prior to starting OKN-007 treatment, whichever is shorter.
3. Patients completing radiotherapy treatment less than 14 days prior to planned study treatment initiation.
4. Current evidence of uncontrolled, significant intercurrent illness that would, in the treating physician's judgment, contraindicate the patient's treatment with OKN-007 due to safety concerns.
5. Patients who, in the opinion of the treating physician, have not fully recovered from recent major surgery to a sufficient extent to tolerate treatment with OKN-007.
6. Known hypersensitivity to OKN-007 or any component in its formulation.
7. Patients taking prohibited medications as described in the current Investigator's Brochure.
8. Patient is pregnant or actively breastfeeding.

Ages: 13 Months to 18 Years | Sex: All
Age Groups: Child, Adult

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Arkansas Children's Research Institute, Little Rock, Arkansas
  - Nicklaus Children's Hospital, Miami, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Children's Hospital and Medical Center, Omaha, Nebraska
  - Prisma Health Midlands Pediatric Hematology/Oncology, Columbia, South Carolina
  - Children's Health, Dallas, Texas
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Carilion Roanoke Memorial Hospital, Roanoke, Virginia